CLINICAL TRIAL: NCT03775681
Title: Is the Gastro LMA a Feasible Alternative to the Use of a Native Airway for Endoscopic Retrograde Cholangiopancreatography (ERCP) Cases?
Brief Title: Feasibility of Laryngeal Mask Airway Gastro on Patients Undergoing Endoscopic Retrograde Cholangiopancreatography for Pancreas and Bile Duct Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0545; NCI-2018-03163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0545 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Bile Duct Disorder; Endocrine Pancreas Disorder
MeSH Terms: conditions — Bile Duct Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde; Interviews as Topic; Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device feasibility (Laryngeal Mask Airway, ERCP) (Experimental): Patients wear Laryngeal Mask Airway after receiving general anesthesia and falling asleep. Patients then undergo standard of care endoscopic retrograde cholangiopancreatography. Patients also complete a 5-minute interview following ERCP procedure.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography; Other: Interview; Device: Laryngeal Mask Airway

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography — Undergo standard of care ERCP
  Other Names: ERCP
Other: Interview — Ancillary studies
Device: Laryngeal Mask Airway — Wear LMA
  Other Names: Laryngeal Mask; LMA

SUMMARY:
This trial determines the feasibility of Laryngeal Mask Airway Gastro (Laryngeal Mask Airway) when used on patients who are undergoing endoscopic retrograde cholangiopancreatography for pancreas and bile duct disorders. Laryngeal Mask Airway is a device that helps patients breathe while they are asleep during procedures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the successful completion of endoscopic retrograde cholangiopancreatography (ERCP) with the Laryngeal Mask Airway (LMA) Gastro.

SECONDARY OBJECTIVES:

I. To determine gastroenterologist satisfaction with the LMA Gastro.

II. To determine anesthesia provider satisfaction with the LMA Gastro.

III. To determine the rate of unsuccessful LMA Gastro placement.

IV. To determine the ability of LMA Gastro to provide adequate oxygenation and ventilation throughout the procedure.

V. To determine and describe the rate of adverse events.

OUTLINE:

Patients wear Laryngeal Mask Airway Gastro after receiving general anesthesia and falling asleep. Patients then undergo standard of care endoscopic retrograde cholangiopancreatography. Patients also complete a 5-minute interview following ERCP procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective ERCP with general anesthesia

Exclusion Criteria:

* Patients with propofol allergy
* Patients at increased aspiration risk
* Patients with abnormal head/neck pathology preventing LMA Gastro placement
* Patients with surgical or radiation treatment to the head/neck making LMA Gastro placement difficult
* Esophagectomy patients
* Patients already intubated upon arrival to endoscopy suite
* Patients undergoing endoscopic ultrasound (EUS)
* Patients with body mass index (BMI) 35 kg/m^2
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hagan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hagan KB, Carlson R, Arnold B, Nguyen L, Lee J, Weston B, Hernandez M, Feng L, Syed T, Hagberg CA. Safety of the LMA(R)Gastro for Endoscopic Retrograde Cholangiopancreatography. Anesth Analg. 2020 Nov;131(5):1566-1572. doi: 10.1213/ANE.0000000000005183. PMID 33079880
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2019 to July 2019
Groups:
- LMA® Gastro™: Upon anesthesia induction, the LMA® Gastro™ was placed in the patient's oropharynx. The cuff was inflated until the cuff pilot indicator line was within the green zone. Appropriate placement was confirmed with end tidal CO2 and adequate tidal volumes of at least 4-5 cc/kg. The LMA® Gastro™ was secured using the manufacturer provided adjustable holder and strap. A standard sideviewing duodenoscope measuring 11.3mm in maximum diameter was lubricated with KY jelly by the gastroenterologist, coating the full length of the endoscope that was inserted into the LMA® Gastro™.
Period: Overall Study
Arm/Group | LMA® Gastro™
Started | 33
Completed | 30
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Race and Ethnicity was not the criteria for Inclusion in the study.
Arm/Group | LMA® Gastro™
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Race and Ethnicity was not the criteria for Inclusion in the study.
  Not Hispanic or Latino | NA — Race and Ethnicity was not the criteria for Inclusion in the study.
  Unknown or Not Reported | NA — Race and Ethnicity was not the criteria for Inclusion in the study.
Region of Enrollment [Number; unit: participants]
  United States | 30
Type of Endoscopic Retrograde Cholangiopancreatography (ERCP) [Count of Participants; unit: Participants] — Type of ERCP cases involving the use of LMA Gastro
  Participants
    Stent Placement | 12
    Stent Removal | 9
    Stent Exchange | 4
    Diagnostic | 3
    Other | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Overall Success of ERCP With LMA Gastro
Description: Successful completion of ERCP with the LMA® Gastro™
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | LMA® Gastro™
Number analyzed (Participants) | 30
Participants | 28

2. Other Pre Specified Outcome: Gastroenterologist and Anesthesiologist Satisfaction With the LMA® Gastro™
Description: Surveys for gastroenterologist and anesthesiologist satisfaction with the Laryngeal Mask Airway (LMA) Gastro contain items measured on a 10-point Likert scale with 1 reflecting strong disagreement and 10 strong agreement. Mean scores and standard deviations will be used to provide summaries for each survey item. Summaries will be stratified by gastroenterologist and anesthesiologist. Paired differences in survey items between gastroenterologist and anesthesiologist scores will be summarized using descriptive statistics and 95% CIs.
Time Frame: Up to 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LMA® Gastro™
Number analyzed (Participants) | 30
score on a scale
  Discordance | 3.45 [0 to 100]
  Concordance | 96.55 [0 to 100]

ADVERSE EVENTS:
Time Frame: Baseline
Description: This is a non-randomized, unblinded feasibility study involving use of LMA Gastro device for ERCP. The device has been deemed low risk and there are no additional risk to the patient. No AE/SAE's to report.
Arm/Group | LMA® Gastro™
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT03775681/Prot_SAP_000.pdf